CLINICAL TRIAL: NCT04630431
Title: Understanding the Challenges, Behavioral Patterns, and Preferences Towards Participation in Clinical Trials in Minority Patient Populations: Development and Validation of a Personalized Clinical Trial Educational Platform to Boost Participation Among Underserved Cancer Patients
Brief Title: Understanding Challenges, Behavioral Patterns, and Preferences Toward Participation in Clinical Trials in Minority Patient Populations: Development of a Personalized Clinical Trial Educational Platform to Increase Participation in Clinical Trials Among Underserved Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MC220901; NCI-2020-08521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-004014 (Other: Mayo Clinic)
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part I (questionnaire, medical record review) (Experimental): Patients complete a questionnaire about their preferences, understanding, and attitudes regarding clinical trials. Patients also have their medical records reviewed.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration
- Part II: Arm A (clinical trial education, standard of care) (Active Comparator): Patients undergo clinical trial education via a video and educational booklet and then standard of care follow-up on study.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Part II: Arm B (clinical trial education, navigation) (Experimental): Patients undergo clinical trial education via a video and educational booklet and then undergo patient navigation with active clinical trial matching and receive clinical trial information through the electronic medical record portal on study.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Electronic Health Record Review; Behavioral: Patient Navigation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo standard of care follow-up
  Other Names: standard of care; standard therapy
  Arms: Part II: Arm A (clinical trial education, standard of care); Part II: Arm B (clinical trial education, navigation)
Other: Educational Intervention — Undergo clinical trial education via a video and educational booklet
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Part II: Arm A (clinical trial education, standard of care); Part II: Arm B (clinical trial education, navigation)
Other: Electronic Health Record Review — Review of medical record
Behavioral: Patient Navigation — Undergo clinical trial navigation
  Other Names: Patient Navigator Program
  Arms: Part II: Arm B (clinical trial education, navigation)
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This clinical trial investigates the challenges, behavioral patterns, and preferences towards participation in clinical trials in minority patient populations in order to develop a personalized clinical trial educational platform to increase participation in clinical trials among underserved cancer patients. Learning more about patients' understanding of clinical trials may help identify barriers that limit patient's participation. Information gathered from this trial will be used to develop educational materials that may aid minority patients in overcoming barriers to participating in clinical trials. A personalized clinical trial educational platform may help increase participation in clinical trials among minority populations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To understand and document patient preferences, understanding, and attitudes regarding clinical trials.

II. To compare patient attitudes regarding clinical trials among cancer patients belonging to different racial/ethnic groups.

III. To establish the magnitude of existing knowledge gap relating to clinical trials among underserved cancer patients and the extent of improvement with a personalized educational approach.

IV. To determine how a personalized educational approach impacts enrollment in clinical trials of underserved cancer patients.

OUTLINE:

PART I: Patients complete a questionnaire about their preferences, understanding, and attitudes regarding clinical trials. Patients also have their medical records reviewed.

PART II: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo clinical trial education via a video and educational booklet and then standard of care follow-up on study.

ARM B: Patients undergo clinical trial education via a video and educational booklet and then undergo patient navigation with active clinical trial matching and receive clinical trial information through the electronic medical record portal on study.

ELIGIBILITY:
Inclusion Criteria:

* PART I: Subjects must be adults with age >= 18 years at the time of study entry
* PART I: Subjects with any cancer diagnosis may be included
* PART I: Subjects must be identified as new patients to hematology oncology at the treating site
* PART I: Subjects must be willing to provide informed consent for the study
* PART II: Subjects must be adults with age >= 18 years at the time of study entry
* PART II: Subjects with any cancer diagnosis may be included
* PART II: Subjects must be identified as new patients to hematology oncology at the treating site
* PART II: Subjects must be willing to provide informed consent for the study

Exclusion Criteria:

* PART I: Patients reported to have an estimated life-expectancy of < 6 months, as assessed by their clinician
* PART I: Patients not willing to complete the Clinical Trials Study survey
* PART II: Patients reported to have an estimated life-expectancy of < 6 months, as assessed by their clinician
* PART II: Patients not willing to complete the education intervention or continued follow up for at least 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Documentation of patient preferences, understanding, and attitudes regarding clinical trials (part I) | Baseline
  Overall percentages of the individual categories for each item of the survey will be summarized across all individuals. Any continuous items collected will be summarized using Means and/or medians depending on the distribution of the data. Most of this analysis will be exploratory and viewed as hypothesis generating.
Comparison of patient attitudes regarding clinical trials among cancer patients belonging to different racial/ethnic groups (part I) | Baseline
  Overall percentages of the individual categories for each item of the survey will be summarized across all individuals. Most of this analysis will be exploratory and viewed as hypothesis generating.
Knowledge score (part II) | Baseline
  Knowledge score at baseline in underserved groups will be compared with knowledge score of non-underserved cancer patients in the study.
Change in knowledge score (part II) | Baseline up to 6 and 12 months
  Knowledge score at baseline will be compared with scores at 6 months and 12 months. Scores of patients enrolled in the educational intervention and in the comparator arm will be reviewed.
Patient enrollment in a clinical trial | Up to 24 months
  The binary outcome of whether or not each patient is enrolled in a trial or not, focusing on the underserved patients. The proportion of patients enrolled in a trial will be compared in each of the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials